CLINICAL TRIAL: NCT06158750
Title: A Prospective, Multicenter, Single Arm Clinical Trial to Evaluate the Safety and Effectiveness of Flow Modulation Device for Intracranial Aneurysms
Brief Title: To Evaluate the Safety and Effectiveness of Flow Modulation Device for Intracranial Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Wallaby Medical Technologies Co.,Inc. (Industry)
Collaborators: Phenox GmbH (Industry); Beijing Wallaby Medical Technologies Co.,Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-1312
Record Dates: First submitted 2023-11-21; First posted 2023-12-06 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): Patients can be included in the study if they meet all of the inclusion and none of the exclusion criteria and have provided written informed consent, intent to use Flow modulation device to treat intracranial aneurysm.
  Interventions: Device: p64/p48 MW HPC Flow Modulation Device

INTERVENTIONS:
Device: p64/p48 MW HPC Flow Modulation Device — Endovascular intervention with p64/p48 MW HPC Flow Modulation Device was performed in patients diagnosed with intracranial aneurysms

SUMMARY:
The purpose of this study is to assess safety and effectiveness of the p64/p48 MW HPC Flow Modulation Device.

DETAILED DESCRIPTION:
Title: A prospective, multicenter, single arm clinical trial to evaluate the safety and effectiveness of Flow Modulation Device for intracranial aneurysms.

Device: p64/p48 MW HPC Flow Modulation Device. Study design: Prospective, multicenter, single arm Clinical Study.

Purpose: To assess safety and effectiveness of p64/p48 MW HPC Flow Modulation Device .

Study duration: 32 months. Sample Size: 120 patients. Number of sites: ≤10. Follow-up time: 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 80 years, male or female;
* Patients diagnosed as intracranial aneurysms by brain CTA/MRA/DSA;
* Patients with unruptured saccular aneurysms or fusiform aneurysm who are clinically determined to use flow modulation device for endovascular treatment;
* The diameter of the target aneurysm parent vessel was 1.75-5mm;
* Patients target aneurysm is planned to be embolized using flow modulation devices only;
* The mRS Score of the patients was 0-2
* Patients understand the purpose of the study, accept the follow-up period, and agree to comply with all requirements, agree to participate in the clinical trial and voluntarily sign the informed consent.

Exclusion Criteria:

* Patients who have contraindications to antiplatelet and/or anticoagulant therapy or do not start antiplatelet therapy in time before treatment;
* Patients with anatomical structure is not suitable for endovascular treatment due to severe vascular tortuosity or stenosis shown by angiography;
* Patients with acute ruptured aneurysm or with a history of intracranial hemorrhage or subarachnoid hemorrhage within 30 days before surgery;
* Patients with target aneurysm treated with endovascular interventional therapy before enrollment;
* Known to be allergic to Nitinol platinum alloy and angiographic agents;
* Conditions that in the opinion of the investigators would prevent patients from completing the study, such as the expected survival period of active tumor less than 1-year, high-risk group of cerebral thrombosis, heart failure and atrial fibrillation;
* The target aneurysms were blood vesicular aneurysms, pseudoaneurysms, or aneurysms associated with arteriovenous malformation, moyamoya disease, or multiple aneurysms that could not be treated by a single flow modulation device;
* Serious infection is not controlled and is not suitable for operation;
* Patients who underwent major surgery or interventional therapy (such as brain, cardiac, chest, abdominal or peripheral vascular) within 30 days before surgery;
* Obvious abnormal coagulation function or bleeding tendency;
* Combined with severe renal insufficiency, creatinine greater than or equal to 200umol/L; Patients with severe liver diseases (such as acute and chronic hepatitis, cirrhosis), or ALT more than 3 times the upper normal limit;
* Pregnancy, lactation, or women of childbearing age who plan to be pregnant during the study period;
* Participation in any other clinical trial within 30 days prior to signing informed consent;
* Other conditions considered by the investigator to be inappropriate for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete occlusion | 12 months
  Raymond grade was evaluated by the independent imaging evaluation Committee 12 months after surgery according to the subjects' imaging results, and the rate of complete aneurysm occlusion was calculated.
  Aneurysm complete occlusion is defined as Raymond Grade I.

SECONDARY OUTCOMES:
Technical success rate | Within 24 hours after surgery
  Technical success is defined as the successful placement of a Flow Modulation Device. Successful implantation means that the Flow Modulation Device is placed at the target site and effectively covers the neck of the aneurysm, and the rest of the device is successfully released and withdrawn to the outside of the body.
Rate of successful occlusion | 6 months, 12 months
  Raymond grade was evaluated by the independent imaging evaluation Committee 6 months and 12 months after surgery according to the subjects' imaging results, and the rate of successful aneurysm occlusion was calculated.
  Aneurysm successful occlusion is defined as Raymond Grade I/II.
Rate of complete occlusion | 6 months
  Raymond grade was evaluated by the independent imaging evaluation Committee 6 months after surgery according to the subjects' imaging results, and the rate of complete aneurysm occlusion was calculated.
  Aneurysm complete occlusion is defined as Raymond Grade I.
Rate of good clinical prognosis | 3 months, 6 months, 12 months
  Good clinical prognosis means mRS 0~2
Rate of in-stent-stenosis | to 6 months, to 12 months
  In-stent-stenosis defined as moderate or severe stenosis of the tumor artery, that is, stenosis > 50%
Device performance evaluation | Within 24 hours after surgery
  After each use of the device, the researchers evaluated the operational performance of the device in terms of conveying, flexibility, compliance and wall adhesion.
Death, stroke, and thrombotic events | to 12 months
  Record the number of death, stroke and thrombotic events throughout the clinical trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Zhang, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No